CLINICAL TRIAL: NCT05434351
Title: A Review on the Clinical Outcome of Chinese Women With Moderate to Severe Symptoms of Genitourinary Syndrome of Menopause (GSM) Treated With Vaginal Dehydroepiandrosterone (DHEA)
Brief Title: The Outcome of Chinese Women With Genitourinary Syndrome of Menopause Treated With Vaginal Dehydroepiandrosterone
Status: Terminated | Type: Observational
Why Stopped: inadequate sample and only few patients were prescribed with vaginal DHEA
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, LAU Yan Yan, Principle investigator, Chinese University of Hong Kong
Other Study IDs: CRE 2022.089
Record Dates: First submitted 2022-05-22; First posted 2022-06-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Genitourinary Syndrome of Menopause
Keywords: vaginal dehydroepiandrosterone (DHEA)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese women with moderate to severe symptoms of genitourinary syndrome of menopause: It is a single-group study.
  Interventions: Other: vaginal dehydroepiandrosterone

INTERVENTIONS:
Other: vaginal dehydroepiandrosterone — the clinical outcome in Chinese women with moderate to severe symptoms of GSM treated with vaginal DHEA for 12 weeks will be evaluated

SUMMARY:
Genitourinary syndrome of menopause (GSM) is a common condition with prevalence was up to 80%. Symptoms associated with GSM include vaginal or vulvar dryness, itchiness, dyspareunia, increased urinary frequency or urgency and dysuria. Although the symptoms are disturbing and causing a significant negative impact on quality of life, it is observed that only a minority of the women receive proper treatment. Treating these GSM-associated symptoms properly is important because these symptoms usually persist with time, unlike vasomotor symptoms of menopause which may subside spontaneously with time.

The clinical efficacy and metabolism of vaginal DHEA has been evaluated in western population. However, there is lack of local data on the effectiveness of vaginal DHEA in treating Chinese women with GSM. Therefore, we aim at evaluating the clinical outcome of our participants who have moderate to severe symptoms of GSM who has been treated with vaginal DHEA.

DETAILED DESCRIPTION:
Genitourinary syndrome of menopause (GSM) is a common condition with prevalence was up to 80%. [1] Symptoms associated with GSM include vaginal or vulvar dryness, itchiness, dyspareunia, increased urinary frequency or urgency and dysuria. [2] Although the symptoms are disturbing and causing a significant negative impact on quality of life, it is observed that only a minority of the women receive proper treatment. Treating these GSM-associated symptoms properly is important because these symptoms usually persist with time, unlike vasomotor symptoms of menopause which may subside spontaneously with time.

Current treatments for GSM-associated symptoms in our unit at Department of Obstetrics and Gynaecology, Prince of Wales Hospital include vaginal moisturizer and local estrogen- based medications. For vaginal moisturizer, they usually fail to alter the underlying pathophysiological change in urogenital tract. For estrogen-containing treatment, long term use is not recommended as systemic absorption of hormones may occur. A new medication, vaginal dehydroepiandrosterone (DHEA) has been introduced to our unit to treat women with moderate to severe symptoms of GSM since July 2021. The clinical efficacy and metabolism of vaginal DHEA has been evaluated in western population. There were four randomized placebo- controlled studies [3-6] showing that 12 weeks treatment of DHEA improved moderate to severe symptoms of GSM. In comparative studies, the efficacy of DHEA was similar to that of conjugated equine estrogen and estradiol. In addition, due to intracrine action of DHEA in particular tissue, it has not showed to increase the level of circulating estrogen or the androgen level beyond the menopausal range. [7]

However, there is lack of local data on the effectiveness of vaginal DHEA in treating Chinese women with GSM. Therefore, we aim at evaluating the clinical outcome of our participants who have moderate to severe symptoms of GSM who has been treated with vaginal DHEA.

All Chinese women who have moderate to severe symptoms of GSM and treated with vaginal DHEA since year 2021-2022. All menopause Chinese women with moderate to severe symptoms of GSM and treated with vaginal DHEA were enrolled for analysis. Menopause is defined as cessation of menses for more than 1 year in women with uterus, or follicle stimulating hormone (FSH) ≥ 40 in women with no menses more than 6 months. Diagnosis of GSM was made after exclusion of other differential diagnosis such as candidiasis / lichen sclerosis/ urodynamic stress incontinence/ detrusor over-activity etc. Moderate to severe symptoms of GSM was defined as a visual analogue score (VAS) of 4 or above of any item including vaginal itchiness, dryness, pain and hotness, dysuria, urinary urgency, stress urinary incontinence, urinary urge incontinence and dyspareunia.

There is a standard dataset for patients presenting with GSM is available in the O&G Department. During the clinic visit, a thorough history and physical examination including abdominal and genital examination will be performed. A transvaginal ultrasound will be performed to determine the endometrial thickness (ET) and exclude other adnexal pathology. Blood taking for hormonal profile was will be performed for baseline check. Mid-stream urinalysis and high vaginal swab will be taken to rule out any infection. After excluding history of hormonal sensitive cancer, active or history of thromboembolic events, unexplained abnormal uterine bleeding and endometrial thickness ≥5mm. If the participant has moderate to severe symptoms of GSM and fit for vaginal DHEA, a 12-week vaginal DHEA will be prescribed. A follow-up appointment will be given in 3-6 months interval to review symptoms. Participants will receive the intervention of vaginal DHEA as a routine medical care.

The medical records of Chinese participants with moderate to severe symptoms of GSM and treated with vaginal DHEA of the aforesaid period will be reviewed. Participant's demographic data, symptoms severity, clinical assessments, investigations, treatment outcome and adverse effect will be collected. The effect of vaginal DHEA will be studied. The end date to the retrospective data collection is 15 Mar 2022.

Genitourinary syndrome of menopause (GSM) is a prevalent but commonly neglected condition. Symptoms can be disturbing to the affected women and affecting their quality of life. The review of the clinical outcome of Chinese women with moderate to severe symptoms of GSM treated with vaginal DHEA allows us to raise awareness of this condition and improve our clinical management. These could also provide a better local evidence of future clinical, research use and patient care.

ELIGIBILITY:
Inclusion Criteria:

• All menopause Chinese women who have moderate to severe symptoms of Genitourinary syndrome of menopause (GSM) and treated with vaginal DHEA

Exclusion Criteria:

* Genitourinary syndrome of menopause (GSM) due to other differential diagnosis such as candidiasis / lichen sclerosis/urodynamic stress incontinence/ detrusor over-activity.
* Amenorrhoea due to medication
* History of hormonal sensitive cancer, active or history of thromboembolic events, unexplained abnormal uterine bleeding
* Endometrial thickness ≥ 5mm

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: All menopause Chinese women with moderate to severe symptoms of GSM and treated with vaginal DHEA were enrolled for analysis.
  Menopause is defined as cessation of menses for more than 1 year in women with uterus, or follicle stimulating hormone (FSH) ≥ 40 in women with no menses more than 6 months.
  Moderate to severe symptoms of GSM was defined as a visual analogue score (VAS) of 4 or above of any item including vaginal itchiness, dryness, pain and hotness, dysuria, urinary urgency, stress urinary incontinence, urinary urge incontinence and dyspareunia.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
The symptoms in Chinese women with moderate to severe symptoms of GSM. | baseline
  The symptoms of GSM were assessed by a visual analogue score (0 to 10) of items including vaginal itchiness, dryness, pain and hotness, dysuria, urinary urgency, stress urinary incontinence, urinary urge incontinence and dyspareunia. The higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The clinical outcome in Chinese women with moderate to severe symptoms of GSM treated with vaginal DHEA | 12-week
  The clinical outcomes were assessed by a visual analogue score (0 to 10) of items including vaginal itchiness, dryness, pain and hotness, dysuria, urinary urgency, stress urinary incontinence, urinary urge incontinence and dyspareunia. The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Yan Lau, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] The NAMS 2020 GSM Position Statement Editorial Panel. The 2020 genitourinary syndrome of menopause position statement of The North American Menopause Society. Menopause. 2020 Sep;27(9):976-992. doi: 10.1097/GME.0000000000001609. PMID 32852449
- [Background] Binkowska M, Paszkowski T, Violetta SP, Wilczak M, Zgliczynski W. Position statement by Experts of the Polish Menopause and Andropause Society, and the Polish Society of Aesthetic and Reconstructive Gynaecology on the medicinal product Intrarosa(R). Prz Menopauzalny. 2019 Dec;18(3):127-132. doi: 10.5114/pm.2019.90113. Epub 2019 Dec 20. No abstract available. PMID 31975978
- [Result] Labrie F, Archer DF, Koltun W, Vachon A, Young D, Frenette L, Portman D, Montesino M, Cote I, Parent J, Lavoie L, Beauregard A, Martel C, Vaillancourt M, Balser J, Moyneur E; VVA Prasterone Research Group. Efficacy of intravaginal dehydroepiandrosterone (DHEA) on moderate to severe dyspareunia and vaginal dryness, symptoms of vulvovaginal atrophy, and of the genitourinary syndrome of menopause. Menopause. 2016 Mar;23(3):243-56. doi: 10.1097/GME.0000000000000571. PMID 26731686
- [Result] Archer DF, Labrie F, Bouchard C, Portman DJ, Koltun W, Cusan L, Labrie C, Cote I, Lavoie L, Martel C, Balser J; VVA Prasterone Group. Treatment of pain at sexual activity (dyspareunia) with intravaginal dehydroepiandrosterone (prasterone). Menopause. 2015 Sep;22(9):950-63. doi: 10.1097/GME.0000000000000428. PMID 25734980
- [Result] Labrie F, Archer DF, Bouchard C, Fortier M, Cusan L, Gomez JL, Girard G, Baron M, Ayotte N, Moreau M, Dube R, Cote I, Labrie C, Lavoie L, Berger L, Gilbert L, Martel C, Balser J. Intravaginal dehydroepiandrosterone (prasterone), a highly efficient treatment of dyspareunia. Climacteric. 2011 Apr;14(2):282-8. doi: 10.3109/13697137.2010.535226. Epub 2011 Jan 18. PMID 21244215
- [Result] Labrie F, Derogatis L, Archer DF, Koltun W, Vachon A, Young D, Frenette L, Portman D, Montesino M, Cote I, Parent J, Lavoie L, Beauregard A, Martel C, Vaillancourt M, Balser J, Moyneur E; Members of the VVA Prasterone Research Group. Effect of Intravaginal Prasterone on Sexual Dysfunction in Postmenopausal Women with Vulvovaginal Atrophy. J Sex Med. 2015 Dec;12(12):2401-12. doi: 10.1111/jsm.13045. Epub 2015 Nov 23. PMID 26597311
- [Result] Labrie F, Cusan L, Gomez JL, Cote I, Berube R, Belanger P, Martel C, Labrie C. Effect of intravaginal DHEA on serum DHEA and eleven of its metabolites in postmenopausal women. J Steroid Biochem Mol Biol. 2008 Sep;111(3-5):178-94. doi: 10.1016/j.jsbmb.2008.06.003. Epub 2008 Jun 12. PMID 18598765